CLINICAL TRIAL: NCT06299618
Title: Environmental Influence on Mental Illness Via Modifications of Genomes and Metabolomes in Adolescents With Autism
Acronym: ENIGMA-I
Status: Not yet recruiting | Type: Observational
Sponsor: University College Cork (Other)
Collaborators: University of Southampton (Other); Carol Davila University of Medicine and Pharmacy (Other); Microlink PC UK LTE (Unknown); Engineering Ingegneria Informatica SpA (Unknown); MEDEA SRL (Unknown); ORTHOKEY ITALIA SRL (Unknown)
Responsible Party: Principal Investigator, Dr. Deirdre Murray, Professor Deirdre Murray, University College Cork
Other Study IDs: ENIGMA-I
Record Dates: First submitted 2023-06-23; First posted 2024-03-08 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Autism; Autism Spectrum Disorder
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to enrich the understanding of the physiological mechanisms that predispose autistic adolescents to mental illness. It will inform a possible pathway and biomarker handprint of mental illness severity and prognosis to formulate a neurobiologically informed personalization strategy that could be applied for selecting appropriate Evidence Based Intervention (EBI) for treating an adolescent formally diagnosed with Autism.

DETAILED DESCRIPTION:
The goal of this observational study is:

1. to identify environmental factors which may significantly contribute to the already vulnerable mental health of autistic adolescents in the age group of 11 - 15 years in developing mental illness;
2. to perform quantitative modelling of the Epigenetic - Genetic/Metabolomic - Mental health (EGM) process chain for designing control strategies based on the subjects' personal, environmental, historical, and current state.

ELIGIBILITY:
Inclusion Criteria:

* Autistic Adolescents
* Must be able to interact verbally
* Parental consent and participants must be able and willing to give written informed assent and to comply with the requirements of the study protocol
* Must be willing to return for all study visits and wear the study device at home
* Must have access to and be able to operate a smartphone.

Exclusion Criteria:

* Adolescents with severe motor impairments or schizophrenia
* Complex medical conditions, which would interfere with ability to take part in the study visits or outcomes.
* Intellectual disability, not capable to attend mainstream school

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be recruited from paediatric and community paediatric clinics. Participants may also be identified through open invitations on websites, social media pages, and through a study specific social media page.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Symptoms of anxiety | Months 0-6
  Symptoms of anxiety will be assessed via the Anxiety Scale for Children (ASC-ASD).
  The ASC-ASD is a 24 item self-report for use with young people aged between 8-16 years with a diagnosis of Autism. Items are rated on a 4-point Likert scale, ranging from 0 to 3. Total score range from 0 to 72, with higher scores indicating higher levels of anxiety. The ASC-ASD will be completed by participants at the clinic visits at month 0, 2, 4, and 6.
Symptoms of anxiety | Months 0-6
  Symptoms of anxiety will be assessed via the Revised Children's Anxiety and Depression Scale-25 (RCADS-25).
  The RCADS-25 is a 25-item self-report, rendering an anxiety subscale with 14 items. Items are scored on a 4-point Likert scale with higher scores representing greater symptom severity. Scores for the anxiety subscale range from 0 to 42. The RCADS-25 will be completed biweekly over the 6-month study duration.
Symptoms of depression | Months 0-6
  Symptoms of depression will be assessed via the Beck Depression Inventory for Youth (BDI-Y).
  The BDI-Y is a 20-item self report. Items are scored on a 4-point Likert scale ranging from 0 to 3. Total scores range from 0 to 60 with higher scores indicating higher symptom severity. The BDI-Y will be completed by participants at the clinic visits at month 0, 2, 4, and 6.
Symptoms of depression | Months 0-6
  Symptoms of depression will be assessed via Revised Children's Anxiety and Depression Scale-25 (RCADS-25).
  The RCADS-25 is a 25-item self-report, rendering a depression subscale with 10 items. Items are scored on a 4-point Likert scale with higher scores representing greater symptom severity. Scores for the depression subscale range from 0 to 30. The RCADS-25 will be completed biweekly over the 6-month study duration.

OTHER OUTCOMES:
Attention-Deficit/Hyperactivity | Months 0-6
  DSM-IV criteria for attention-deficit/hyperactivity disorder (ADHD) will be assessed using the SNAP-IV 18-item scale, an abbreviated version of the Swanson, Nolan, and Pelham (SNAP) Questionnaire. Items are rated on a 4-point Likert scale with higher scores indicating higher symptom levels. The two subsets of symptoms pertain to Inattention (items 1-9) and Hyperactivity/Impulsivity (items 10-18), with possible scores ranging from 0 to 27 for each subset. The SNAP-IV will be completed by participants' parents within 72 hours prior to the at clinic visits at months 0, 2, 4, and 6.
Sleep disturbance | Months 0-6
  Sleep disturbance will be assessed using the Sleep Disturbance Scale for Children (SDSC), consisting of 26 items, rated on a 5-point Likert scale. The total score ranges from 26-130 with higher scores indicating higher levels of sleep disturbance. Besides the total score, 6 subscales representing more specific sleep disturbance will be calculated, i.e., difficulty in initiating and maintaining sleep (DIMS); sleep breathing disorders (SBD); disorders of arousal (DoA); sleep-wake transition disorders (SWTD); disorders of excessive somnolence (DOES); sleep hyperhidrosis (SH). The SDSC will be completed by participants' parents within 72 hours prior to the at clinic visits at months 0, 2, 4, and 6.
Physical Activity | Months 0-6
  Levels of physical activity over the past week will be assessed using the Physical Activity Questionnaire for Older Children (PAQ-C). The PAQ-C consists of 10-items, with items 1-9 being rated on 5-point Likert scales, scored from 1-5. The overall activity summary score is represented by the mean of items 1-9, thus ranging from 1 to 5, with higher scores indicating higher levels of physical activity. The PAQ-C will be completed by participants within 72 hours prior to the at clinic visits at months 0, 2, 4, and 6.
Symptoms of Mental Health Disorders | Month 0 and Month 6
  Mental health disorder symptoms will be assessed via the Development and Well-Being Assessment (DAWBA), an online questionnaire/interview package indicating likely DSM-5 psychiatric diagnoses. Participants and parents will complete the online questionnaires within 72 hours prior to Visit 1 and Visit 4. The DAWBA covers Separation anxiety, Specific phobia, Social phobia, Panic disorder / agoraphobia, Post-traumatic stress disorder, Obsessive compulsive disorder, Generalised anxiety disorder, Body dysmorphic disorder, Disruptive mood dysregulation disorder, Major depression, ADHD / hyperkinesis, Oppositional defiant disorder, Conduct disorder, Eating disorders, including anorexia, bulimia and binge eating, Autism spectrum disorders, Tic disorders, including Tourette syndrome, Bipolar disorders. Diagnostic predictions are given at probability bands, i.e., (1) less than 0.1% (--), (2) around 0.5% (-), (3) around 3% (+/-), (4) around 15% (+), (5) around 50% (++), (6) above 70% (+++).
Cognitive Assessment | Month 0 and Month 6
  Cognitive assessment will be conducted using the Cambridge Neuropsychological Test Automated Battery (CANTAB), a cognitive assessment research software, administered via a touchscreen device. The battery for participants with a diagnosis of Autism consists of measures examining executive functions, planning, episodic memory, and processing speed. CANTAB is language independent and requires no prior familiarity with computers. It will be administered at clinic during Visit 1 and Visit 4.
Nutritional Assessment | Months 0-6
  Nutritional assessment is based on an adapted version of the Nutritional Assessment for Children and Adults with ASD (NACA-ASD). The NACA-ASD was designed to assist families and researchers in making a rough estimate of the quality of diet and nutritional supplementation of a person with Autism. Participants will be asked to estimate the number of servings of different food groups they have eaten over the past 24 hours. Assessment will be conducted at clinic during all visits.
Heart Rate | Months 0-6
  Heart Rate in Beats per Minute (BPM) will be assessed via the noninvasive Vivalink wearable electrocardiogram (ECG) patch (ECG sampling 128 Hz; Heart rate range 40-300 BPM). Participants will be asked to wear the sensor for 5 days in the first 2 weeks following the baseline visit (i.e., 10 days total). Subsequently, they will be asked to wear the sensor for 72 hours every other week over the study course.
Respiratory Rate | Months 0-6
  Respiratory rate will be assessed via the noninvasive Vivalink wearable electrocardiogram (ECG) patch. It is collected in Breaths per Minute (BrPM) with a range of 5 to 25 BrPM. Participants will be asked to wear the sensor for 5 days in the first 2 weeks following the baseline visit (i.e., 10 days total). Subsequently, they will be asked to wear the sensor for 72 hours every other week over the study course.
Genotype | Month 0
  Infinium Global Screening Array-24 BeadChip with DNA from buccal swab at visit 1 will be utilised. Bead array content is selected for imputation accuracy at minor allele frequencies of >1% across Genomes Project populations. Clinical research content includes variants with established disease associations, relevant pharmacogenomics markers, and curated exonic content based on databases. After intensity calling, sample quality control includes removing samples with genotyping call rate <98% and SNPs with a call rate <98% or Hardy-Weinberg equilibrium p-value <5 × 10-6. For imputation, array-derived genotypes were prephased using SHAPEITv2 and imputation was carried out using IMPUTE2 software with 1000 Genomes phase 3 reference panel. SNPs with minor allele frequency <.10 and an IMPUTE2 'info' matric <.9 were excluded to ensure max. confidence in imputation quality. Each SNP will be coded 0,1,2; associations with environmental factors and mental health will be examined.
DNA Methylation | Months 0-6
  DNA methylation will be assessed using the Illumina Infinium MethylationEPIC v2.0 BeadChip array from DNA extracted from buccal swabs collected at each visit. The EPIC array is a genome-wide methylation screening tool that targets over 935,000 CpG sites in the most biologically significant regions of the human methylome. Infinium 850K data will be processed using the Bioconductor package minfi in R (version 3.4.2). Beta-mixture quantile (BMIQ) normalization will be used to remove array biases and correct for probe design. DNA methyaltion will be a continous measures with values between 0 and 1. Robust regression models using limma will be run to assess associations between DNA methylation and the measured environmental factors, genotype and mental health outcomes together with changes in DNA methylation over time.
Hormone Levels | Months 0-6
  Hormone levels in urine will be assessed using ELISAs and Mass spectrometry from samples taken at each visit. These methods will give ug/ml measures of the different hormones assessed. Hormone levels will then be compared to the measured environmental parameters, DNA methylation, metabolome, and mental health outcomes.
Metabolomic Profile | Months 0-6
  Metabolic profiles of urine and faecal samples will be measured by nuclear magnetic resonance (NMR) spectroscopy (700 MHz Bruker spectrometer equipped with a cryoprobe and autosampler) and liquid-chromatography-mass spectrometry (LCMS) (Waters Premier LC system hyphenated to a Waters Synapt Q-TOF). These approaches will be applied in an untargeted manner to measure a broad range of biochemical classes (e.g., amino acids, sugars, organic acids, vitamins, aromatic compounds). Multivariate metabolic profiles will be processed and analysed using bespoke pipelines in Matlab and R. Statistical approaches used will include, but will not be limited to, principal components analysis, projection to latent structures, self-organising maps, DIABLO, and random forests. These methods will be employed to highlight metabolite features and data structures related to mental health, environmental parameters, DNA methylation and genotype data.

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Murray, PhD, Principal Investigator — University College Cork, Cork, Ireland; Geraldine Boylan, PhD, Principal Investigator — University College Cork, Cork, Ireland; Mihai Berteanu, PhD, Principal Investigator — University of Medicine and Pharmacy, Bucharest, Romania; Samuele Cortese, PhD, Principal Investigator — University of Southampton, Southampton, UK; Koushik Maharatna, PhD, Principal Investigator — University of Southampton, Southampton, UK
Locations (3):
- University College Cork, Cork, Ireland
- University of Medicine and Pharmacy Carol Davila Bucharest, Bucharest, Romania
- University of Southampton, Southampton, United Kingdom